CLINICAL TRIAL: NCT01964313
Title: Comprehensive Intervention and Outcome Research Programs for Acute Coronary Syndrome
Brief Title: Acute Coronary Syndrome Genetic Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University First Hospital (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Yong Huo, Director, Department of Cardiology, Peking University First Hospital
Other Study IDs: 2011BAI11B06
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; treatment strategy; genetics
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 4ml of vein blood are to be retained for genetic analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ACS cohort: Patients diagnosed with acute coronary syndrome.

SUMMARY:
To describe the role of genetic factors and its relationship and interaction with environmental factors in the recurrence of cardiac events in Chinese patients with acute coronary syndrome.

DETAILED DESCRIPTION:
* Research cohort: Patients diagnosed with acute coronary syndrome are enrolled and to be followed up for 2 years.
* Baseline and follow up variables include patients' demographics, medical history, ACS event characteristics, clinical treatment options (interventional cardiology, drug therapy: antithrombotic therapy, other treatments recommended by guidelines ) and follow up events information.
* Blood Sample collection 4ml of vein blood will be drawed. Centrifugation of plasma and WBC will be done on-site within 30 minutes for DNA extraction. Samples will be stored at -80℃ freezer for subsequent applications.
* A nested case-controlled study is designed for the genetic analysis:

  1. Cases: Patients suffered from death, myocardial infarction, stroke and coronary revascularization and bleeding during the 2-year follow up. We expected to get 600 cases in the study cohort;
  2. Controls: among patients without any of the above events during follow, matched controls of 1:1 ratio will be selected according to date of admission (± 1 month), age (± 5 years), sex, baseline ACS diagnosis, whether treated with PCI , the same pattern of antithrombotic therapy and the study center.
* Genotyping Genotype testing using exome DNA chips (Exome Beadchip). Exome Beadchip is a high-throughput DNA chip designed by Illumina's, containing 240,000 SNP on exons in the genome that may lead to functional changes.
* Analysis:

  1. To analysis the impact of genetic characteristics on selection of treatment strategy in ACS patients, and its interaction with other baseline clinical variables.
  2. To analysis the impact of genetic characteristics on patient outcomes, and its interaction with clinical characteristics and management patterns.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been provided.
* Contact Order Form has been provided.
* Aged 18 years or older.
* Diagnosis of STEMI, NSTEMI or UA using the following definitions:

  1. Criteria for STEMI diagnosis:

     1. History of chest pain/discomfort and
     2. Persistent ST-segment elevation (> 30 min) of ≥ 0.1 mV in 2 or more contiguous ECG leads or presumed new left bundle branch block (LBBB) on admission and
     3. Elevation of cardiac biomarkers (CK-MB, troponins): at least one value above the 99th percentile of the local laboratory upper reference limit.
  2. Criteria for NSTEMI diagnosis:

     1. History of chest pain/discomfort and
     2. Lack of persistent ST-segment elevation, LBBB or intraventricular conduction disturbances and
     3. Elevation of cardiac biomarkers (CK-MB, troponins): at least one value above the 99th percentile of the local laboratory upper reference limit.
  3. Criteria for Unstable Angina diagnosis:

     1. Symptoms of angina at rest or on minimal exercise and
     2. At least 0.5mm ST deviation in at least 2 leads and
     3. No increase in biomarkers of necrosis
     4. OR objective evidence of ischaemia by non-invasive imaging OR significant coronary stenosis as determined by the treating physician at angiography if this is standard practice in study site.
* Hospitalized within 48 hours of onset of symptoms.

Exclusion Criteria:

Patients will not be eligible to participate if any of the following exclusion criteria are present:

* UA, STEMI and NSTEMI precipitated by or as a complication of surgery, trauma, or GI bleeding or post-PCI.
* UA, STEMI and NSTEMI occurring in patients already hospitalized for other reasons.
* Presence of any condition/circumstance which in the opinion of the investigator could significantly limit the complete follow up of the patient (e.g. tourist, non-native speaker or does not understand the local language, psychiatric disturbances).
* Presence of serious/severe co-morbidities in the opinion of the investigator which may limit short term (i.e. 6 month) life expectancy.
* Current participation in a randomised interventional clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from 75 hospitals in China.
Sampling Method: Non-Probability Sample
Enrollment: 3422 (Estimated)
Dates: Start 2012-07; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events | 2 year
  Death, Myocardial infarction, stroke, coronary revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First hospital, Beijing, Beijing Municipality, China